CLINICAL TRIAL: NCT02577783
Title: Doxorubicin Hydrochloride Liposome vs Doxorubicin Combined With Bortizomib and Dexamethasone to Treat Initially Diagnosed Multiple Myeloma: A Randomized Prospective Clinical Study
Brief Title: PDD vs PAD to Treat Initially Diagnosed MM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ5202
Record Dates: First submitted 2015-10-07; First posted 2015-10-16 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: Doxorubicin Hydrochloride
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDD arm (Experimental): patients involved in PDD arm will accept chemotherapy of PDD regimen (doxorubicin hydrochloride liposome plus bortizomib and dexamethasone )
  Interventions: Drug: PDD regimen: doxorubicin hydrochloride iposome, bortizomib and dexamethasone
- PAD arm (Active Comparator): patients involved in PAD arm will accept chemotherapy of PAD regimen (doxorubicinplus bortizomib and dexamethasone )
  Interventions: Drug: PAD regimen: bortizomib, dexamethasone and doxorubicin

INTERVENTIONS:
Drug: PDD regimen: doxorubicin hydrochloride iposome, bortizomib and dexamethasone — doxorubicin hydrochloride iposome (duomeisu) plus bortizomib (velcade) and dexamethasone (disaimisong)
  Arms: PDD arm
Drug: PAD regimen: bortizomib, dexamethasone and doxorubicin — doxorubicin (duoroubixing) plus bortizomib (velcade) and dexamethasone (disaimisong)
  Arms: PAD arm

SUMMARY:
The purpose of this study is to determine whether doxorubicin hydrochloride liposome is superior to doxorubicin when combined with bortizomib and dexamethasone for treating patient with initially diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and untreated multiple myeloma patients
* Patients with age between 18 and 70 years
* With a evaluable disease
* ECOG score ≤2
* NE≥1.0×10E9 /L, Plt≥50×10E9 /L, Hb≥70 g/L
* AST, ALT, ALP≤3×ULN, serum BIL≤ULN
* LVEF≥ 50%
* Not in pregnancy
* Written informed consent are acquired

Exclusion Criteria:

* Severe heart failure (NYHA grade II or higher)
* Active and uncontrolled severe infection
* HIV positive
* Have accepted any other anti-tumor drug within 30 days before the first dose of doxorubicin hydrochloride iposome or doxorubicin
* Grade 2 or higher peripheral neuropathy before treatment
* Have suffered any other malignancy in past 5 years
* Females in lactation
* Other situations that investigators consider as contra-indication for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-10; Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 4 cycles (each cycle is 28 days) of chemotherapy
  sCR + CR + VGPR

SECONDARY OUTCOMES:
Overall remission rate | 4 cycles (each cycle is 28 days) of chemotherapy
  sCR + CR
Progression-free survival | 3 year
Adverse Event | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China